CLINICAL TRIAL: NCT03180983
Title: Effect of a Nurse-centered Multimodal Intervention on Prescribing Antibiotics in Nursing Home: A Randomized Cluster Study
Brief Title: Antibiotic Use in French Nursing Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Paris 13 (Other)
Responsible Party: Principal Investigator, Monique ROTHAN-TONDEUR, Head of nursing research chair, University of Paris 13
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Prot_ATOUM4_V1; NCT03994523 (obsolete NCT alias)
Record Dates: First submitted 2017-06-01; First posted 2017-06-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Antibiotic Resistant Infection

STUDY DESIGN:
Intervention Model Description: CLUSTER RANDOMIZED STUDY
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTIONAL GROUP (Other): The intervention group will receive a blended-learning intervention.
  Interventions: Behavioral: multimodal intervention
- CONTROL GROUP (No Intervention): No intervention

INTERVENTIONS:
Behavioral: multimodal intervention — Investigators will propose an online training. In addition, investigators will make phone calls to nursing home interlocutor between two nursing home visits. The tools of this intervention will consist on posters , quiz about bacteriuria and urinary tract infection (UTI) and algorithm to help nurse's reasoning when UTI is suspected.
  Arms: INTERVENTIONAL GROUP

SUMMARY:
CONTEXT: France is still one of the biggest consumers of antibiotics in Europe. An explanation for this increase in consumption would be aging. Thus, part of this aging population lives in nursing home, where the urinary tract infection is the second most suspected pathology. However, it can most often be bacteriuria requiring no antibiotic therapy. In nursing home, nurses who alert prescribers when an infection is suspected by describing clinical signs.However, his propensity to perform too rapidly and systematically an examination with dipsticks leads the physician to prescribe antibiotic. This is how a program called ATOUM is set up to reduce the prescription of antibiotics in nursing home. The present ATOUM 4 study builds on this program.

OBJECTIVE: To measure the effect of a nurse-centered multimodal intervention involving training and sensitization on urinary tract infection, asymptomatic bacteriuria, antibiotic resistance and interprofessional communication on antibiotic therapy. METHODS: This will be a randomized double-arm interventional study in 40 nursing home. The intervention group of 20 nursing home will receive a blended-learning intervention.

DETAILED DESCRIPTION:
CONTEXT: France is still one of the biggest consumers of antibiotics in Europe. An explanation for this increase in consumption would be aging. Thus, part of this aging population lives in nursing home, where the urinary tract infection is the second most suspected pathology. However, it can most often be bacteriuria requiring no antibiotic therapy. In nursing home, nurses alert prescribers when an infection is suspected by describing clinical signs. However, their propensity to perform too rapidly and systematically an examination with dipsticks leads physicians to prescribe antibiotic. This is how a program called ATOUM is set up to reduce the prescription of antibiotics in nursing home. The present ATOUM 4 study builds on this program.

OBJECTIVE: To measure the effect of a nurse-centered multimodal intervention involving training and sensitization on urinary tract infection, asymptomatic bacteriuria, antibiotic resistance and interprofessional communication on antibiotic therapy. METHODS: This will be a randomized double-arm interventional study in 40 nursing home. The intervention group of 20 nursing home will receive a blended-learning intervention.The primary outcome will be the percentage of reduction in antibiotic prescription at the end of the twelve months following the first visit to nursing home. This data, aggregated by nursing home, will be obtained from the structures concerned via their prescription registration system.

ELIGIBILITY:
Inclusion Criteria:

* nursing home with registred nursing
* Presence of prescription registration system
* Situated in Paris and surb of Paris

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Antibiotics prescription for UTI | Twelve months
  The percentage of reduction in prescriptions of antibiotics for urinary tract infection

SECONDARY OUTCOMES:
Total prescriptions of antibiotics | Twelve months
  whatever the infection

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franchi C, Tettamanti M, Pasina L, Djignefa CD, Fortino I, Bortolotti A, Merlino L, Nobili A. Changes in drug prescribing to Italian community-dwelling elderly people: the EPIFARM-Elderly Project 2000-2010. Eur J Clin Pharmacol. 2014 Apr;70(4):437-43. doi: 10.1007/s00228-013-1621-6. Epub 2014 Jan 8. PMID 24398968
- [Background] Moreira VG, Lourenco RA. Prevalence and factors associated with frailty in an older population from the city of Rio de Janeiro, Brazil: the FIBRA-RJ Study. Clinics (Sao Paulo). 2013 Jul;68(7):979-85. doi: 10.6061/clinics/2013(07)15. PMID 23917663
- [Background] Smith PW, Bennett G, Bradley S, Drinka P, Lautenbach E, Marx J, Mody L, Nicolle L, Stevenson K; Society for Healthcare Epidemiology of America (SHEA); Association for Professionals in Infection Control and Epidemiology (APIC). SHEA/APIC Guideline: Infection prevention and control in the long-term care facility. Am J Infect Control. 2008 Sep;36(7):504-35. doi: 10.1016/j.ajic.2008.06.001. No abstract available. PMID 18786461
- [Background] Smith PW, Bennett G, Bradley S, Drinka P, Lautenbach E, Marx J, Mody L, Nicolle L, Stevenson K; SHEA; APIC. SHEA/APIC guideline: infection prevention and control in the long-term care facility, July 2008. Infect Control Hosp Epidemiol. 2008 Sep;29(9):785-814. doi: 10.1086/592416. No abstract available. PMID 18767983
- [Background] Marston HD, Dixon DM, Knisely JM, Palmore TN, Fauci AS. Antimicrobial Resistance. JAMA. 2016 Sep 20;316(11):1193-1204. doi: 10.1001/jama.2016.11764. PMID 27654605
- [Background] Phillips CD, Adepoju O, Stone N, Moudouni DK, Nwaiwu O, Zhao H, Frentzel E, Mehr D, Garfinkel S. Asymptomatic bacteriuria, antibiotic use, and suspected urinary tract infections in four nursing homes. BMC Geriatr. 2012 Nov 23;12:73. doi: 10.1186/1471-2318-12-73. PMID 23176555
- [Background] Chami K, Gavazzi G, Carrat F, de Wazieres B, Lejeune B, Piette F, Rothan-Tondeur M. Burden of infections among 44,869 elderly in nursing homes: a cross-sectional cluster nationwide survey. J Hosp Infect. 2011 Nov;79(3):254-9. doi: 10.1016/j.jhin.2011.08.003. Epub 2011 Sep 6. PMID 21899920
- [Background] Inkster T, Marek A, Khanna N. Improving antimicrobial prescribing by targeting clinical nurse practitioners. J Hosp Infect. 2010 Sep;76(1):85-6. doi: 10.1016/j.jhin.2010.05.009. No abstract available. PMID 20663586
- See also: Related Info — https://www.ined.fr/fr/tout-savoir-population/chiffres/france/structure-population/population-sexe-ages/
- See also: Related Info — https://www.google.com/search?q=%C3%89volution+2000-2010+de+la+consommation+d%E2%80%99antibiotiques+en+France&ie=utf-8&oe=utf-8
- See also: Related Info — http://www.insee.fr/fr/themes/tableau.asp?reg_id=20&ref_id=santc06108
- See also: Related Info — http://www.insee.fr/fr/publications-et-services/sommaire.asp?ref_id=TEF15